CLINICAL TRIAL: NCT03534752
Title: Clinical Characteristics of Adult Patients With Inborn Errors of Metabolism in French-speaking Switzerland
Brief Title: Retrospective Study of Adult Patients With Inborn Errors of Metabolism in Switzerland
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Christel Tran, Principal Investigator, University of Lausanne
Other Study IDs: 2017-02328
Record Dates: First submitted 2018-04-10; First posted 2018-05-23 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Inborn Errors of Metabolism
Keywords: Inborn errors of Metabolism; Adulthood; Clinical characteristics
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study aimed at establishing a database of the current health of adult patients with IEM in the French-speaking part of Switzerland. .

DETAILED DESCRIPTION:
Background Inborn errors of metabolism (IEMs) are a group of rare disorders caused by genetic mutations that affect enzymes of intermediary metabolism. Because adult with IEMs has become an emerging and challenging group in Switzerland, this study is intended to assess the actual situation of adult patients with IEM in the French-speaking part of Switzerland, namely their age, their sex, their diagnosis, age at disease onset and their clinical outcome including complications of the disease.

All adult patients with a biochemical and/or genetic diagnosis of IEM followed at the adult metabolic clinic from the Lausanne University Hospital and Geneva University Hospital between 01.10.2013 to 31.12.2017 will be included in the study. In addition, investigators will also include the patients referred to the clinic for suspicion of IEM and determinate if the investigation confirmed an IEM disease. Electronic and paper patient charts will be reviewed for clinical features, biochemical investigations, molecular genetic testing, diagnostic imaging, treatment and long-term outcome. All data will be entered in an Excel database.

ELIGIBILITY:
Inclusion Criteria:

* All IEM adult patients who were transitioned from the pediatric clinic to the adult metabolic clinic (the Centre for Molecular Disease in Lausanne and the Division of Endocrinology, Diabetology, Hypertension and Nutrition of the HUG) since its creation in 2013 and those who were referred to our clinic for suspicion of IEM and requiring further investigation.

Exclusion Criteria:

* Age < 16 years . Any document attesting a refusal to participate will exclude the data entry of the concerned patient.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient clinic for Adult patients with Inborn Errors of Metabolism from the Lausanne University Hospital (Division of Genetic Medicine) and Geneva University Hospital (Division of Endocrinology, Diabetology, Hypertension and Nutrition of the HUG.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Specific diagnosis of IEM listed by their frequency | First visit
  Clinical outcome
Age at diagnosis (years/months) | First visit
  Clinical outcome
Medical complications | 4 years
  Clinical outcome including acute liver failure, nephropathy, metabolic acidosis, ophthalmologic anomalies, epilepsy, encephalopathy, myopathy, neuropathy, diabetes
Specific treatment for Inborn Errors of Metabolism | 4 years
  Treatment specific to each diseases including ammonia scavenger, enzyme replacement therapy, carnitine, ubiquinone, vitamins, specific diet, dialysis, specific metabolic formula
Number of hospital admission | 4 years
  Clinical outcome
Survival rate (%) | 4 years
  Clinical Outcome
Gender (Male/female) | First visit
  Demography outcome

SECONDARY OUTCOMES:
Abdominal Ultrasound results | 4 years
  Radiological Imaging description of spleen and/or liver when available (size, echostructure)
Magnetic resonance Imaging scan | 4 years
  Radiological Imaging description of brain, abdomen and bone when available
Bone density test | 4 years
  Radiological Imaging description of bone including T-score when available
Biological biomarkers of specific diseases (lysosomal storage disorders and galactosemia) | 4 years
  Laboratory including blood concentration of chitotriosidase and Galactose-1-Phosphate
Clinical chemistry | 4 years
  Laboratory including blood concentration of sodium, potassium, liver function tests, creatinine, uric acid, urea, amino acids, acylcarnitine profile, methylmalonate, total homocysteine and urine concentration of organic acids
Hematology tests | 4 years
  Laboratory (blood count, international normalized ratio, prothrombin time)
Enzyme activity in leucocytes and/or fibroblasts | 4 years
  Enzyme activity of deficient enzyme when available for lysosomal storage diseases, mucopolysaccharidoses, cobalamin deficiency, diseases, classical homocystinuria
Molecular analysis results of candidate gene for Inborn Errors of metabolism | 4 years
  Laboratory including mutation results confirming the molecular origin of the disease when available

OTHER OUTCOMES:
Educational level | 4 years
  Demography outcome
Profession | 4 years
  Demography outcome

CONTACTS AND LOCATIONS:
Overall Officials: Christel Tran, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospitals, Lausanne, Canton of Vaud, Switzerland